CLINICAL TRIAL: NCT04182308
Title: Anatomic Characteristics of Lisfranc Ligament in Vietnamese Adult
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Nguyen Phu Chan, Orthopeadic resident, clinical physician, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: IRB00010195
Record Dates: First submitted 2019-11-24; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Lisfranc Injury
MeSH Terms: interventions — Dissection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: dissection — Dissection of lisfranc ligament from 30 aldult Vietnamese cadavers's foot

SUMMARY:
Goal: the aim of this study is to determine the anatomic characteristic of lisfranc ligament

DETAILED DESCRIPTION:
Goal: the aim of this study is to determine the anatomic characteristic of lisfranc ligament, including components, thickness, height, and width, origins as well as relationship of center point of origin with neighbor structures in Vietnamese adults

ELIGIBILITY:
Inclusion Criteria:

* above ankle amputation samples at Cho Ray hospital, HCM city, Vietnam

Exclusion Criteria:

* foot injuries
* foot infection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: above ankle amputation samples at Cho Ray hospital, HCM city, Vietnam
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Some anatomic characteristic of lisfranc ligament | 2 years
  lenght, width

SECONDARY OUTCOMES:
relative position with neighbor structures | 2 years
  cm

CONTACTS AND LOCATIONS:
Overall Officials: Hung P Do, professor, Study Director — Cho Ray Hospital
Locations (1):
- Cho Ray hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
not yet

REFERENCES:
- [Result] Johnson A, Hill K, Ward J, Ficke J. Anatomy of the lisfranc ligament. Foot Ankle Spec. 2008 Feb;1(1):19-23. doi: 10.1177/1938640007312300.. PMID 19825687